CLINICAL TRIAL: NCT04370223
Title: A Trial of Ozone Auto-hemotherapy in Adults Hospitalized With Covid-19 Pneumonia
Brief Title: Ozone Auto-hemotherapy for COVID-19 Pneumonia
Acronym: COVID-OZONE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Collaborators: Clinica Nuestra Senora del Rosario (Other)
Responsible Party: Principal Investigator, Marc Vives, MD, PhD, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 Networking group
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19 Pneumonia
Keywords: Ozone therapy; Covid-19; SARS-COV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone auto-hemotherapy plus standard treatment (Experimental): Patients in the ozone auto-hemotherapy group will receive treatment mixing 100-200ml of blood with ozone at a concentration of 40 μg / mL with a gas volume of 200 ml. Treatment will occur every 12h during 5 days.
  Interventions: Biological: Ozone auto-hemotherapy
- Standard treatment alone (No Intervention): Standard treatment will be the one used in each hospital participating in the trial.

INTERVENTIONS:
Biological: Ozone auto-hemotherapy — ozone auto-hemotherapy
  Arms: Ozone auto-hemotherapy plus standard treatment

SUMMARY:
This is a multicenter, randomized, controlled, open-label clinical trial testing the use of ozone auto-hemotherapy in hospitalized patients with Covid-19 pneumonia.

Eligible patients will be randomly assigned to receive either ozone auto-hemotherapy plus standard treatment, or standard treatment alone.

Patients in the ozone auto-hemotherapy group will receive treatment mixing 100-200ml of blood with ozone at a concentration of 40 μg / mL with a gas volume of 200 ml. Treatment will occur every 12h during 5 days. Standard treatment will be the one used in each hospital participating in the trial.

All analyses will be done according to the intention-to-treat principle

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 confirmed by positive polymerase chain reaction (PCR) for Severe Acute Respiratory Syndrome (SARS-COV-2) in respiratory tract sample, plus pneumonia confirmed by imaging tests and arterial oxygen saturation (SpO2) <94% with ambient air or a partial pressure of oxygen to fraction of inspired oxygen (pO2/FiO2) ratio <300 mmHg or SpO2/FiO2 ≤ 315.
* Acceptance to participate in the study and signing of the informed consent.

Exclusion Criteria:

* Patients who have received treatment with any form of ozone therapy 6 months before admission to the hospital.
* Patients who have previously been treated and have experienced some type of adverse reaction to ozone therapy.
* Patients aware of having a deficiency of Glucose-6-phosphate dehydrogenase.
* Patients with clinically decompensated chronic comorbidities, independently of COVID-19.
* Patients suffering from any psychiatric disorder specified in axis I of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V), other than major depression.
* Patients who are not able to clearly understand the objectives and methodology of the study.
* Pregnant or lactating patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-10-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Rate of patients achieving improvement in clinical condition at day 14 after recruitment | 14 days
  Improved clinical condition defined by an improvement of 2 points in the clinical status, 8 categories, ordinary score of the World Health Organization (WHO)

SECONDARY OUTCOMES:
Mortality at day 28 | 28 days
  mortality
Rate of patients achieving improvement in clinical condition at day 28 after recruitment | 28 days
  Improved clinical condition defined by an improvement of 2 points in the clinical status, 8 categories, ordinary score of the World Health Organization (WHO)
Rate of patients achieving improvement in clinical condition at day 7 after recruitment | 7 days
  Improved clinical condition defined by an improvement of 2 points in the clinical status, 8 categories, ordinary score of the World Health Organization (WHO)
Time to clinical improvement or hospital discharge | 28 days
  Improved clinical condition defined by an improvement of 2 points in the clinical status, 8 categories, ordinary score of the World Health Organization (WHO)
Number of ventilator-free days at 28 days | 28 days
  Ventilator-free days from last extubation day until day 28 after recruitment
Hospital length of stay | 28 days
  Days hospitalized
Time to a 2-fold decrease in ferritin | 14 days
  Number of days until a 2-fold decrease in ferritin (ng/mL)
Time to a 2-fold decrease in C-protein reactive | 14 days
  Number of days until a 2-fold decrease in C-Protein Reactive (mg/L)
Time to a 2-fold decrease in Dimer-D | 14 days
  Number of days until a 2-fold decrease in Dimer-D (ng/mL)
Time to a 2-fold decrease in Lactate Dehydrogenase | 14 days
  Number of days until a 2-fold decrease in Lactate Dehydrogenase (U/L)
Time to a 2-fold decrease in Neutrophils to Lymphocytes ratio | 14 days
  Number of days until a 2-fold decrease in Neutrophils to Lymphocytes ratio

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Universitari Dr Josep Trueta, Girona
  - Clinica Nuestra Señora del Rosario, Ibiza Town
  - Hospital Quirón Rey Juan Carlos I, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Príncipe de Asturias de Alcalá de Henares, Madrid
  - Fundació Althaia de Manresa, Manresa
  - Hospital Vithas Valencia Consuelo, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Clinica Claro, Vigo

IPD SHARING:
Plan to Share IPD: No